CLINICAL TRIAL: NCT04008940
Title: A Retrospective Radiological Analysis of the Mechanical Performance of Different Locking Plates in Distal Femoral Fractures
Brief Title: Locking Plates for Distal Femur Fractures - a Multicenter Case Review
Acronym: VA_LCP
Status: Completed | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: VA_LCP
Record Dates: First submitted 2019-04-17; First posted 2019-07-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Distal Femur Fracture
Keywords: VA-LCP DF; LCP DF; LISS DF; various angle locking plate
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Distal femur plates — By assessing the rate and mode of mechanical failures we aim to identify risk factors for mechanical failures among the analysed plate types. This, finally, is depending on the overall number of cases and number of failure cases.

SUMMARY:
In order to assess the rate and mode of failure cases observed in patients with distal femur fractures treated with a distal femur plates, anonymized radiographs from those patients will be collected retrospectively.

All available images will reviewed by an expert review board in regards to fracture classification, implant and surgery details, quality of initial reduction and plate positioning as well as the occurrence of mechanical complications and the outcome in terms of fracture healing (if available). Additionally, age and gender as basic demographical data will be collected in a de-identified way..

DETAILED DESCRIPTION:
Severely comminuted distal femur fractures can be challenging injuries and usually require surgical treatment with lateral distal plate osteosynthesis.

Anatomically pre-contoured locking plates are commonly used. In 2012, the 4.5mm VA-LCP Curved Condylar Plate for distal femur fractures (VA-LCP DF, Synthes) was introduced offering the option of axis variation of the locking screws.

Recently, a report highlighted cases of implant failure with this implant, cautioning practicing surgeons against the use of this implant in certain type of AO/OTA fracture and dislocation classification 33 fractures (AO/OTA classification).

Based on this report, the current study was designed to perform a retrospective in-depth radiological analysis of all cases distal femur fractures of 4 participating sites in which the VA-LCP DF, the LCP Distal Femur Plate (LCP DF, Synthes) or the 'less invasive stabilization system' for distal femur fractures (LISS DF, Synthes) were used for fracture stabilization. The radiological in-depth analysis will be done by an expert review board with the aim to identify potential causes and risk factors for the failure cases among all cases collected.

This evaluation will contribute to a better understanding of the mechanical performance of distal femur fracture plates and the causes and risk factors for failures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of a distal femur fracture type OTA/AO classification 33-A, -B, -C
* uni- or bilateral
* low or high energy trauma
* Open or closed fractures
* Surgical treatment with the VA-LCP DF, LISS DF, LCP DF
* Available radiographical documentation, beginning with the injury radiographs, ending with the documented healing or any documented failure with or without revision surgery (up to a maximum follow-up of 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age 18 years and older
  * Diagnosis of a distal femur fracture type OTA/AO classification 33-A, -B, -C
  * uni- or bilateral
  * low or high energy trauma
  * Open or closed fractures
  * Surgical treatment with the VA-LCP DF, LISS DF, LCP DF
  * Available radiographical documentation, beginning with the injury radiographs, ending with the documented healing or any documented failure with or without revision surgery (up to a maximum follow-up of 1 year
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Fracture | baseline
  type of fracture
Fracture classification | baseline
  AO/OTA classification 33A, -B or C
Mechanism of injury | baseline
  High energy trauma (H) or low energy trauma assessed as H for high and L for low energy trauma
Implant used | baseline
  Implant manufacturer name (VA-LCP DF, LISS DF, LCP DF)
Open or closed fracture | 1 year
  G-A class: Y=open, N=closed
Bone union in time | baseline until 1 year
  weeks to bone union

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lee, MD, Principal Investigator — University of California Davis, Dept. of Orthopaedic Surgery
Locations (5):
- United States (3):
  - University of California, Sacramento, California
  - Houston, Texas
  - Inova Orthopedics, Fairfax, Virginia
- Switzerland (2):
  - Kantonsspital Liestal, Liestal, Basel-Landschaft
  - Kantonsspital Graubünden, Chur, Kanton Graubünden

IPD SHARING:
Plan to Share IPD: No